CLINICAL TRIAL: NCT03192943
Title: A Phase 1 Study for Safety and Tolerability of BMS-986205 Administered in Combination With Nivolumab (BMS-936558) in Advanced Malignant Tumors
Brief Title: A Study of BMS-986205 Given in Combination With Nivolumab in Patients With Advanced Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA017-048
Record Dates: First submitted 2017-06-14; First posted 2017-06-20 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — linrodostat; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dose Escalation (Experimental): monotherapy and combination therapy
  Interventions: Drug: BMS-986205; Biological: Nivolumab

INTERVENTIONS:
Drug: BMS-986205 — Specified dose on specified days
Biological: Nivolumab — Specified dose on specified day
  Other Names: Opdivo; BMS-936558

SUMMARY:
The purpose of this study is to assess the safety and tolerability for the combination therapy of BMS-986205 and Nivolumab in patients with advanced tumors

ELIGIBILITY:
Inclusion Criteria:

For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

* Participants must have histologic or cytological confirmation of a malignancy that is advanced (metastatic and/or unresectable) with measureable disease per Response Evaluation Criteria In Solid Tumors (RECIST v1.1)
* Participants must have received, and then progressed or been intolerant to standard treatment regimen in the advanced or metastatic setting
* Eastern Cooperative Oncology Group performance status of ≤ 1

Exclusion Criteria:

* Participants with known or suspected CNS metastases, untreated CNS metastases, or with the CNS as the only site of disease are excluded
* History of congenital or autoimmune hemolytic disorders
* History or presence of hypersensitivity or idiosyncratic reaction to methylene blue

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | 15 months
  Safety and Tolerability
Incidence of Serious Adverse Events (SAEs) | 15 months
  Safety and Tolerability
Incidence of Death | 15 months
  Safety and Tolerability
Incidence of Laboratory Abnormalities | 15 months
  Safety and Tolerability
AEs leading to discontinuation | Up to one year
  Safety and Tolerability

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to one year
  To characterize the Pharmacokinetics (PK) of BMS-986205 administered alone and in combination with nivolumab
Time of maximum observed plasma concentration (Tmax) | Up to one year
  To characterize the PK of BMS-986205 administered alone and in combination with nivolumab
Area under the plasma concentration-time curve in one dosing interval [AUC(TAU)] | Up to one year
  To characterize the PK of BMS-986205 administered alone and in combination with nivolumab
Trough observed plasma concentration at the end of the dosing interval (Ctrough) | Up to one year
  To characterize the PK of BMS-986205 administered alone and in combination with nivolumab
Apparent total body clearance (CLT/F) | Up to one year
  To characterize the PK of BMS-986205 administered alone and in combination with nivolumab
Apparent volume of distribution at steady-state (Vss/F) | Up to one year
  To characterize the PK of BMS-986205 administered alone and in combination with nivolumab
Percent urinary recovery over 24 hours (%UR24) | Up to 24 hours
  To characterize the PK of BMS-986205 administered alone and in combination with nivolumab
Biomarker Availability | Up to one year
  To characterize the pharmacodynamic activity of BMS-986205 administered alone and in combination with nivolumab
Incidence of anti-drug antibody (ADA) | Up to one year
  To characterize the immunogenicity of nivolumab when administered in combination with BMS-986205
Best Overall Response (BOR) | Up to one year
  To investigate the preliminary anti-tumor activity of BMS-986205 administered in combination with nivolumab in advanced malignant tumors
Duration of Response (DOR) | Up to one year
  To investigate the preliminary anti-tumor activity of BMS-986205 administered in combination with nivolumab in advanced malignant tumors

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Chuo-ku, Tokyo, Japan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm